CLINICAL TRIAL: NCT01804764
Title: Educational and Organizational Intervention's Effect on Severe Sepsis and Septic Shock Management Out of Intensive Care Units: Medical Wards and Emergency Departments
Brief Title: Lotta Alla Sepsi Ospedaliera - Fighting Hospital Sepsis
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: IX/001137-23/12/2010
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Severe Sepsis
Keywords: Severe Sepsis; Septic Shock; Sepsis Six bundle
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sepsis is widespread (1.8 million cases annually worldwide) and accounts for a very high mortality: 20-25% of all severe sepsis, 40-70% of all septic shock. The Surviving Sepsis Campaign (SSC) recommends a first 6 hours "resuscitative bundle" to improve patient's outcome. Despite this, the bundle is poorly performed, because of a superficial knowledge of the guidelines and several difficulties in their clinical implementation. In recognition of this, a "sepsis six" bundle is designed to facilitate early intervention with just three diagnostic and three therapeutic steps to be delivered by staff within 1 h.

The aim of our study is to evaluate if an Educational and Organizational Intervention (EOI) could improve septic patient's outcome in no Critical Care Units. The second endpoint is to evaluate if the compliance to the "sepsis six" bundle could improve after this sort of intervention.

DETAILED DESCRIPTION:
Methods 39 Medical Wards and 12 Emergency Departments, belonging to 12 hospitals, were voluntarily enrolled. Through the collaboration of 12 Multidisciplinary Teams (MT), we took a Pre-EOI picture of the human resources (i.e. doctors to patients ratio) and of the organisational structures (i.e. laboratory's opening hours) of each hospital. For six months, each unit enrolled was asked to fill in a Clinical Checklist for every patient suspected for severe sepsis or septic shock; so that the Pre-EOI "sepsis six" bundle compliance could be evaluated. Then, we planned several pre-agreed educational meetings for all of the doctors and nurses belonging to the enrolled wards. In the meanwhile the MT worked to overcome any impediment to a better septic patient management. Finally, the educated medical staff was asked to fill in again the same Clinical Checklist used in the Pre-EOI phase; so that the Post-EOI "sepsis six" bundle compliance could be evaluated and a comparison with the Pre-EOI phase could be done.

Hypothesis This is the first study aimed to analyze the impact of an Educational and Organizational Intervention in the outcome of septic patients managed in no Critical Care Units. We guess that the differences showed in human resources and organizational structures among the hospitals could have a role in the "sepsis six" bundle compliance and in the patient's outcome, but only a comparison with data collected from the clinical checklist and patient's outcome will confirm our guess. Likewise, we believe that an educational intervention could improve the septic patient's management, but we need the Post-EOI phase conclusion to demonstrate or not our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Any patient having a SIRS due to Sepsis and at least on of the following criteria: Systolic Blood Pressure < 90 mmHg and/or serum lactate > 4 mg/dl and/or organ failure

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the Emergency Department out-patients and the Medical Wards in -patients presenting with suspected svere sepsis or septic shock
Sampling Method: Non-Probability Sample
Enrollment: 1123 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
An improvement in Sepsis Six Bundle implementation for Severe Sepsis and Septic Shock | within 12 months after an Educational and Organizational Intervention

SECONDARY OUTCOMES:
All cause Mortality | 1 month afte diagnosis of Severe Sepsis / Septic Shock

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Vesconi, MD, Study Director — Niguarda Ca' Granda Hospital
Locations (1):
- Niguarda Ca' Granda Hospital, Milan, Italy

REFERENCES:
- [Background] Cardoso T, Carneiro AH, Ribeiro O, Teixeira-Pinto A, Costa-Pereira A. Reducing mortality in severe sepsis with the implementation of a core 6-hour bundle: results from the Portuguese community-acquired sepsis study (SACiUCI study). Crit Care. 2010;14(3):R83. doi: 10.1186/cc9008. Epub 2010 May 10. PMID 20459716
- [Background] Micek ST, Roubinian N, Heuring T, Bode M, Williams J, Harrison C, Murphy T, Prentice D, Ruoff BE, Kollef MH. Before-after study of a standardized hospital order set for the management of septic shock. Crit Care Med. 2006 Nov;34(11):2707-13. doi: 10.1097/01.CCM.0000241151.25426.D7. PMID 16943733
- [Background] Thiel SW, Asghar MF, Micek ST, Reichley RM, Doherty JA, Kollef MH. Hospital-wide impact of a standardized order set for the management of bacteremic severe sepsis. Crit Care Med. 2009 Mar;37(3):819-24. doi: 10.1097/CCM.0b013e318196206b. PMID 19237883
- [Background] Funk D, Sebat F, Kumar A. A systems approach to the early recognition and rapid administration of best practice therapy in sepsis and septic shock. Curr Opin Crit Care. 2009 Aug;15(4):301-7. doi: 10.1097/MCC.0b013e32832e3825. PMID 19561493
- [Background] Girardis M, Rinaldi L, Donno L, Marietta M, Codeluppi M, Marchegiano P, Venturelli C; Sopravvivere alla Sepsi Group of the Modena-University Hospital. Effects on management and outcome of severe sepsis and septic shock patients admitted to the intensive care unit after implementation of a sepsis program: a pilot study. Crit Care. 2009;13(5):R143. doi: 10.1186/cc8029. Epub 2009 Sep 3. PMID 19728879
- [Background] Cronshaw HL, Daniels R, Bleetman A, Joynes E, Sheils M. Impact of the Surviving Sepsis Campaign on the recognition and management of severe sepsis in the emergency department: are we failing? Emerg Med J. 2011 Aug;28(8):670-5. doi: 10.1136/emj.2009.089581. Epub 2010 Jul 26. PMID 20660901
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Talan DA, Moran GJ, Abrahamian FM. Severe sepsis and septic shock in the emergency department. Infect Dis Clin North Am. 2008 Mar;22(1):1-31, v. doi: 10.1016/j.idc.2007.09.005. PMID 18295681
- [Background] Ferrer R, Artigas A, Levy MM, Blanco J, Gonzalez-Diaz G, Garnacho-Montero J, Ibanez J, Palencia E, Quintana M, de la Torre-Prados MV; Edusepsis Study Group. Improvement in process of care and outcome after a multicenter severe sepsis educational program in Spain. JAMA. 2008 May 21;299(19):2294-303. doi: 10.1001/jama.299.19.2294. PMID 18492971
- See also: Surviving Sepsis Campaign Guidelines — http://www.survivingsepsis.org